CLINICAL TRIAL: NCT06161753
Title: The Costs and Effectiveness of Cognitive Functional Therapy for People with Persistent Low Back Pain, Multi-morbidity and Affected by Health Inequality: a Primary Care Mixed Methods Cohort Study.
Brief Title: The Costs and Effectiveness of Cognitive Functional Therapy for People with Persistent Low Back Pain in Coventry.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN634623
Record Dates: First submitted 2023-11-28; First posted 2023-12-08 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain
Keywords: low back pain; population health management; cognitive functional therapy; health inequality
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: mixed-methods single cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Functional Therapy (Experimental): The Cognitive Functional Therapy arm will be subject to receiving the intervention, as described in the intervention section.
  Interventions: Behavioral: Cognitive Functional Therapy

INTERVENTIONS:
Behavioral: Cognitive Functional Therapy — CFT is an individualised, combined physical and behavioural approach specifically developed to target the multidimensional complexity of persistent LBP. CFT utilises a multidimensional clinical reasoning framework that enables the clinician to identify both modifiable and non-modifiable biopsychosocial factors (i.e. physical, cognitive, emotional, social, lifestyle and health comorbidities) underlying an individual's LBP. CFT targets these factors by: (1) helping the patient 'make sense of their pain' from a biopsychosocial perspective, (2) build confidence to engage in valued activities through functional movement training and (3) adopt positive lifestyle behaviours (O'Sullivan et al., 2018).
  Participants will receive approximately 7 treatment sessions over a 13-week period, although this will vary depending on participant needs, in line with the individualised nature of the intervention. Participants will be provided a booster session at 26 weeks to reinforce self-management.
  Other Names: CFT

SUMMARY:
Previous studies have shown Cognitive Functional Therapy (CFT) results in sustained clinically important improvements compared to a variety of interventions for persistent low back pain (LBP). However, CFT is yet to be evaluated in people with persistent LBP who are affected by health inequality and multimorbidity despite the strong association between LBP, socioeconimic deprivation, multimorbidity, and increased prevalance in people from minority ethnic backgrounds. This study will aim to examine the cost and effectiveness of CFT in a population living with LBP, adversely affected by health inequality and multimorbidity in areas of social deprivation in Coventry, United Kingdom.

DETAILED DESCRIPTION:
This study will be conducted in two phases. In Phase 1, a single cohort study will be conducted, whereby Cognitive Functional Therapy (CFT) will be delivered to 150 participants recruited from the physiotherapy waiting list.

Healthcare utilisation data will be collected retrospectively from participants electronic health records and the physiotherapy referral information for the 13 weeks before the date of enrolment. Clinical outcomes will be collected at baseline prior to participants beginning the intervention. Both healthcare utilisation and clinical outcomes will be collected on two further occasions, at 13 and 26 weeks. CFT will be delivered by six physiotherapists who have undergone a comprehensive training programme and demonstrated ability to deliver the intervention to a competency standard, assessed by a CFT tutor using a predefined competency framework used in previous CFT studies. Treatment fidelity will be assessed throughout the study.

In Phase 2, qualitative semi-structured interviews and/or dyad interviews will be conducted with at least 10 participants and their treating physiotherapist. This aims to explore the experiences and acceptability of the intervention for people from this population, the intervention training and the study of participants and physiotherapists.

ELIGIBILITY:
Inclusion Criteria:

* Documented LBP for more than three months.
* Over 18 years old.
* Currently not working - either unemployed or in receipt of long-term sickness benefits at time of enrolment on the study.
* Living in 20% most deprived area of Coventry as defined by Index of Multiple Deprivation (IMD).
* Documented physical and/or mental health co-morbidities (e.g., anxiety, depression, obesity, diabetes, cardiovascular disease).
* Prescribed medications not currently recommended for LBP by NICE Guidelines - opioids, selective serotonin reuptake inhibitors, tricyclic antidepressants, antidepressants and/or gabapentinoids (NICE, 2020).
* Ability to provide informed consent.

Exclusion Criteria:

* Lack capacity, or unable, to provide informed consent.
* Have signs and/or symptoms of serious spinal pathology (less than 2% of all people with LBP (Hartvisgen et al., 2018)) e.g., fracture, infection, acute loss of lower limb motor control, symptoms of cauda equina syndrome or cancer, acute inflammatory disease (e.g. ankylosing spondylitis).
* Have any medical condition that prevents from being physically active.
* Are currently pregnant or are three months post-partum.
* Are unable or unwilling to travel to CoCHC for the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of Healthcare consultations | Baseline (for preceding 13 weeks); 13 weeks; 26 weeks
  Number of healthcare contacts
Prescribed medications, including dosage and frequency | Baseline (for preceding 13 weeks); 13 weeks; 26 weeks
  Prescription medications, dosage and frequency
Imaging requests | Baseline (for preceding 13 weeks); 13 weeks; 26 weeks
  Requests for diagnostic imaging / work-up
Referrals into secondary care | Baseline (for preceding 13 weeks); 13 weeks; 26 weeks
  Referrals made into secondary care (e.g. Orthopaedics, Neurosurgery, Pain Clinic)
Work status | Baseline (for preceding 13 weeks); 13 weeks; 26 weeks
  Work status
Quality Adjusted Life Years | Baselines; 13 weeks; 26 weeks
  Quality Adjusted Life Years will be calculated using the EuroQol 5 Dimensions, 5 level version (EQ5D-5L) and the EuroQol Visual Analogue Scale (EQ-VAS), measure of health-related quality of life.
  The EQ5D-5L consists of five dimensions where the participant indicates their health state by ticking the box next to the most appropriate statement in each of the five dimensions from 1 (lowest impact) to 5 (highest impact). The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ-VAS requires the participant to score their overall health from 0 (worst health imaginable) to 100 (best health imaginable).

SECONDARY OUTCOMES:
Roland-Morris Disability Questionnaire (RMDQ) | Baseline; 13 weeks; 26 weeks
  Activity limitation and disability will be measured using the RMDQ. The RMDQ consists of 24 statements related to disability and activities of daily living. Respondents tick each statement that applies to them at the time of completion, giving a score between 0 (no disability) and 24 (maximum disability).
Numerical Pain Rating Scale (NPRS) | Baseline; 13 weeks; 26 weeks
  Pain intensity will be measured using the Numerical Pain Rating Scale (NPRS). The NPRS asks a person to rate their pain intensity, on average over the previous week, on a scale of 0-10 (11 possible responses), where 0 implies 'no pain at all' and 10 is equal to 'pain as bad as you can imagine'.
Treatment Satisfaction | 13 weeks; 26 weeks
  Participant satisfaction with their allocated intervention will be measured using a simple satisfaction questionnaire containing four responses to the question "how satisfied were you with the care you received for your low back pain? 'Very dissatisfied', 'dissatisfied', 'neither satisfied or dissatisfied', 'satisfied' and 'very satisfied'.
Work Ability Index (WAI) | Baseline; 13 weeks; 26 weeks
  Perceived ability to work will be measured using the Work Ability Index (WAI). The WAI asks a person to rate their current ability to work on a scale of 0-10 (11 possible responses), where 0 implies 'Currently cannot work at all' and 10 is equal to 'Work ability at its best'.
Patient Acceptable Symptoms State (PASS) | Baseline; 13 weeks; 26 weeks
  Perceived level of symptom acceptability will be measured using the Patient Acceptable Symptoms State (PASS). The PASS asks the participant to answer a simple 'Yes' or 'No' answer to the question "Taking into account all of the activities you have during your daily life, your levels of pain, and also your functional impairment, do you consider that your current state is satisfactory?"

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Newton, Principal Investigator — University Hospitals Coventry and Warwickshire NHS Trust
Locations (1):
- City of Coventry Health Centre, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: No